CLINICAL TRIAL: NCT06937528
Title: Knee Osteoarthrosis (KOA) in Jordanian Patients: a Phase I Dose-finding Study Using Extracellular Vesicles (EV) for Advanced Stage III and IV KOA
Brief Title: Use of Extracellular Vesicles (EV) for Knee Osteoarthrosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Abdalla Awidi Abbadi, MD (Unknown); The University of Jordan (Unknown)
Responsible Party: Principal Investigator, Hanan Jafar, Principal Investigator, University of Jordan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVKneeUJCTC
Record Dates: First submitted 2024-02-27; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthrosis
Keywords: osteoarthrosis; Knee; Extracellular vesicles
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extracellular vesicles (EV) (Experimental): Intra-articular Extracellular vesicles injection will be given to each patient in 2 doses
  Interventions: Biological: Extracellular vesicles

INTERVENTIONS:
Biological: Extracellular vesicles — Intra-articular extravascular vesicles injection.
  Other Names: EV

SUMMARY:
Extracellular vesicles (EV) will be injected in patients diagnosed with Knee osteoarthrosis

DETAILED DESCRIPTION:
50 patients from both genders diagnosed with Knee osteoarthrosis, will be enrolled according to strict inclusion and exclusion criteria. These patients will be injected with Extracellular vesicles (EV). Then, they are followed by clinical assessment, laboratory investigations as well as magnetic resonance imaging (MRI) of the injected knee.

ELIGIBILITY:
Inclusion Criteria:

* Severe KOA stage III or IV by Laurance & Kellgren staging as judged by Posterioranterior (PA) Xray of the knee joint.
* Willing to participate by signing the informed consent

Exclusion Criteria:

* Sublaxation beyond 20 degrees of the bones of the knee joint
* Oral anticoagulants or heparin therapy
* Heart failure or arrhythmia
* Body Mass Index > 35
* Uncontrolled Diabetes Mellitus.
* Evidence of Infectious Diseases.
* Active infection
* Malignancy
* Pregnancy
* Anemia less than 11g/dl or thrombocytopenia less than 100,000 or leucopenia less than 3000.
* Unreliable patients
* Non-resident in Jordan

Ages: 42 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety | follow-up duration is 12 months
  Measuring and evaluating the Safety and Tolerability of the intra-articular injection of extracellular vesicles:
  Complete Blood Count (CBC):
  Hemoglobin (Hb) Hematocrit (Hct) White blood cells (WBCs) Platelets (PLTs) Red blood cell indices (MCV, MCH, MCHC) A. Liver Function Tests (LFTs) Alanine aminotransferase (ALT) Asparate aminotransferase (AST) Alkaline phosphatase (ALP) Gamma-glutamyl transferase (GGT) Total bilirubin (TBIL), Direct & Indirect bilirubin Albumin and total protein B. Kidney Function Tests Blood Urea Nitrogen (BUN) Serum Creatinine Uric Acid Estimated Glomerular Filtration Rate (eGFR) C. Electrolyte Panel Sodium (Na⁺) Potassium (K⁺) Calcium (Ca²⁺) Magnesium (Mg²⁺) Chloride (Cl-) Bicarbonate (HCO₃-) D. Glucose & Lipid Profile Fasting blood glucose (FBG) Total cholesterol, HDL, LDL, Triglycerides Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) INR (International Normalized Ratio)

SECONDARY OUTCOMES:
Efficacy | follow-up duration is 12 months
  Measuring and evaluating the efficacy of the Intra Articular Injection of extracellular vesicles measure pain score by questionnaire: KOOS (Knee Injury and Osteoarthritis Outcome Score) Extension of WOMAC, more detailed
  Domains:
  Pain
  Symptoms
  Activities of daily living (ADL)
  Sport and recreation
  Quality of life (QoL)
  Scoring: 0-100 scale (0 = extreme symptoms, 100 = no symptoms)
  Use: Young and active OA patients, post-surgery (e.g., ACL, TKA)

CONTACTS AND LOCATIONS:
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No